CLINICAL TRIAL: NCT01167569
Title: Double-Blind, Randomized Study of High Dose Vitamin C On Outcome in Cardiac Surgery Patients
Brief Title: Study of High Dose Vitamin C On Outcome in Cardiac Surgery Patients
Acronym: VitaminC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 0220070054
Record Dates: First submitted 2010-02-05; First posted 2010-07-22 (Estimated); Results first posted 2020-10-19 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-09

CONDITIONS: Reperfusion Injury
Keywords: Free Radicals; Ascorbic Acid; Cardiac Surgery; Prevention of Reperfusion Injury
MeSH Terms: conditions — Reperfusion Injury | interventions — Ascorbic Acid; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- A-Ascorbic Acid (Vitamin C) (Active Comparator): Ascorbic Acid (Vitamin C) 10mg/kg x 2 in the operating room followed by Ascorbic Acid (Vitamin C) 5mg/kg every 4 hours x 48 hours.
  Interventions: Drug: Ascorbic Acid
- B-5% Dextrose Water or Normal Saline (Placebo Comparator): 5% Dextrose Water or Normal Saline (placebo) x 2 in the operating room followed by 5 % Dextrose Water or NS (placebo) every 4 hours X 48 hours.
  Interventions: Other: 5 % Dextrose Water or Normal Saline

INTERVENTIONS:
Drug: Ascorbic Acid — Ascorbic Acid/Placebo 10mg/kg body weight X2 in Operating Room followed by Ascorbic Acid/Placebo 5mg/kg x 48 hours.
  Other Names: Vitamin C
  Arms: A-Ascorbic Acid (Vitamin C)
Other: 5 % Dextrose Water or Normal Saline — 100 ml D5W or NS X 2 in operating room and then every 4 hours for 48 hours.
  Other Names: D5W or NS
  Arms: B-5% Dextrose Water or Normal Saline

SUMMARY:
It has been shown that the stress that occurs during cardiac surgery leads to early decrease of many of the body's resources such as Vitamin C (ascorbic acid) which may contribute to complications after surgery.

This study will investigate the effects of high doses of intravenous (IV) Vitamin C on the outcome and complications after cardiac surgery.

DETAILED DESCRIPTION:
Patients undergoing cardiac surgery are at significant risk for multiple major complications beyond those associated with other major operations. Most patients survive these events, but up to 10% develop injury to organ systems including the kidneys, lungs, pancreas, brain, etc. It has been shown that the stress that occurs during this critical period (cardiac surgery) leads to early decrease of many of the body's resources such as Vitamin C (ascorbic acid) which seem to contribute to these complications.

This study will investigate the effects of high doses of intravenous (IV) Vitamin C administered before, during and after the cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients 18 years or older undergoing elective or urgent (prior to hospital discharge) cardiac surgery.

Exclusion Criteria:

* History of renal insufficiency, nephrolithiasis, G6PD (glucose-6-phosphate dehydrogenase deficiency) or the chronic use of steroids.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2007-10; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alan Spotnitz, Principal Investigator — Rutgers RWJMS
Locations (1):
- Robert Wood Johnson University Hospital, New Brunswick, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from Oct. 31, 2007 thru July 22, 2009 in the Cardiothoracic Surgery Clinic.
Groups:
- A-Ascorbic Acid (Vitamin C): Ascorbic Acid
  Ascorbic Acid: Ascorbic Acid/Placebo 10mg/kg body weight X2 in Operating Room followed by Ascorbic Acid/Placebo 5mg/kg every 4 hours x 48 hours.
- B-5% Dextrose Water or Normal Saline (Placebo: 5% Dextrose Water or Normal Saline (placebo)
  5 % Dextrose Water or Normal Saline: 100 ml D5W or NS X 2 in operating room and then every 4 hours for 48 hours.
Period: Overall Study
Arm/Group | A-Ascorbic Acid (Vitamin C) | B-5% Dextrose Water or Normal Saline (Placebo
Started | 28 | 29
Completed | 27 | 27
Not Completed | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- A-Ascorbic Acid (Vitamin C): Ascorbic Acid
  Ascorbic Acid: Ascorbic Acid/Placebo 10mg/kg body weight X2 in Operating Room followed by Ascorbic Acid/Placebo 5mg/kg x 48 hours.
- B-Placebo: 5% Dextrose Water or Normal Saline (placebo)
  5 % Dextrose Water or Normal Saline: 100 ml D5W or NS X 2 in operating room and then every 4 hours for 48 hours.
- Total: Total of all reporting groups
Arm/Group | A-Ascorbic Acid (Vitamin C) | B-Placebo | Total
Number analyzed (Participants) | 28 | 29 | 57
Age, Continuous [Mean (Standard Deviation); unit: years] | 69 (2) | 65 (2) | 67 (2)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 17 | 29
  >=65 years | 16 | 12 | 28
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 6 | 13
  Male | 21 | 23 | 44
Region of Enrollment [Number; unit: participants]
  United States | 28 | 29 | 57

OUTCOME MEASURES:

1. Primary Outcome: Mortality
Description: Number of patients who expire within 30 days of their surgery (both in patients and discharged patients)
Time Frame: 30 days
Measure: Number; unit: participants
Groups:
- B-Placebo: 5% Dextrose Water or Normal Saline (placebo) x 2 in the operating room followed by 5 % Dextrose Water or NS (placebo) every 4 hours X 48 hours.
  5 % Dextrose Water or Normal Saline: 100 ml D5W or NS X 2 in operating room and then every 4 hours for 48 hours.
Arm/Group | A-Ascorbic Acid (Vitamin C) | B-Placebo
Number analyzed (Participants) | 28 | 29
participants | 0 | 0

2. Secondary Outcome: Renal Insufficiency
Description: The number of patients who develop renal insufficiency during hospitalization.
Time Frame: hospital discharge
Population: The PI has left the institution, all efforts to locate the data have been exhausted and therefore no results are available to be reported"
Arm/Group | A-Ascorbic Acid (Vitamin C) | B-5% Dextrose Water or Normal Saline (Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | A-Ascorbic Acid (Vitamin C) | B-5% Dextrose Water or Normal Saline
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/29
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/29
Other Adverse Events (participants affected / at risk) | 0/28 | 0/29

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No